CLINICAL TRIAL: NCT04699552
Title: Effect of Laser Settings on Postoperative Voiding Symptoms in Patients Undergoing Holmium Laser Enucleation of the Prostate: A Randomized Prospective Trial
Brief Title: Effect of Laser Settings on Postoperative Voiding Symptoms in Patients Undergoing Holmium Laser Enucleation of the Prostate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI does not wish to move forward with the Study
Sponsor: Indiana University (Other)
Collaborators: Lumenis Be Ltd. (Industry)
Responsible Party: Principal Investigator, Marcelino Rivera, Assistant Professor of Urology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2010195334
Record Dates: First submitted 2021-01-05; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Prostate Disease; Surgery
Keywords: Holmium Laser Enucleation; Prostate
MeSH Terms: conditions — Prostatic Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Treating surgeons will know the randomization at the time of the operation however the postoperative data analysis and results will be performed by the research team in a blinded fashion when examining clinical outcomes and adverse events
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- 2J 20 Hz (Experimental): The power settings of 2J of energy will be consistent between the three treatment arms. The frequency will be 20Hz
  Interventions: Device: 120W Lumenis Holmium:YAG laser 20J
- 2J 40 Hz (Experimental): The power settings of 2J of energy will be consistent between the three treatment arms. The frequency will be 40Hz
  Interventions: Device: 120W Lumenis Holmium:YAG laser 40 J
- 2J 60 Hz (Experimental): The power settings of 2J of energy will be consistent between the three treatment arms. The frequency will be 60Hz
  Interventions: Device: 120W Lumenis Holmium:YAG laser 60 J

INTERVENTIONS:
Device: 120W Lumenis Holmium:YAG laser 20J — 120W Lumenis Holmium:YAG laser 20J
  Arms: 2J 20 Hz
Device: 120W Lumenis Holmium:YAG laser 40 J — 120W Lumenis Holmium:YAG laser 40J
  Arms: 2J 40 Hz
Device: 120W Lumenis Holmium:YAG laser 60 J — 120W Lumenis Holmium:YAG laser 60J
  Arms: 2J 60 Hz

SUMMARY:
The purpose of this study is to evaluate the safety and outcomes, such as postoperative dysuria (pain during urination), urgency (frequent need to urinate) and urinary incontinence (leaking urine or inability to hold urine), of 3 different HoLEP laser settings.

DETAILED DESCRIPTION:
Study subjects will be identified by the clinical team or study coordinator either at the time surgery is scheduled or by review of the surgery schedule. Each subject will be screened for inclusion/exclusion criteria by reviewing the chart. If inclusion/exclusion criteria are met, the patient will be approached by a member of the research team for enrollment into the study. The patient must consent to participate by reviewing a study-specific, IRB-approved informed consent form before any study data is collected.

After informed consent has been obtained, a complete medical history including a detailed urologic history will be obtained prior to the HoLEP procedure. Standard pre-operative laboratory tests will be obtained, including a complete blood count, basic metabolic panel and urine culture.

Pre-operative, intra-operative and post-operative management of the patients included in this study will not differ from routine HoLEP treatment options described in the literature and practiced at our center. All laser settings examined are currently utilized. A complete description of the HoLEP procedure at our institution has previously been described15. Briefly, a 550um Lumenis MOSES fiber will be utilized. A 120W Holmium:YAG laser made by Lumenis will be used. Operatively, the time (minutes) for resection of the tissue will be recorded as "enucleation time". Once enucleation of the tissue has been completed, the time (in minutes) for complete removal of the enucleated tissue will be recorded as "morcellation time". Enucleated tissue can be removed by any means determined necessary by the surgeon, i.e. he/she may use the holmium laser or graspers in combination with the morcellator. Enucleation is typically performed in a stepwise fashion with an initial groove at the 5 and 7 o'clock position, followed by enucleation of the median lobe. The enucleation of the lateral lobes occurs in a bottom up approach. At times depending on patient anatomy an intraoperative decision by the treating surgeon may result in an early apical release. The power settings of 2J of energy will be consistent between the three treatment arms. The frequency will differ from 20Hz, 40Hz and 60Hz between the three treatment arms. After enucleation, hemostasis is performed at a setting of 1J and 20 Hz with a widened pulse width for standard HoLEPs. For patients with a high median bar of bladder neck tissue, a single incision at the bladder neck is made at 6 o'clock. Total amount of laser energy utilized for the procedure will also be recorded.

Note will be made of concurrent procedures done at the time of HoLEP including: bladder calculi managed with cystolithopaxy or upper urinary tract calculi management.

Postoperative, patients will be provided with daily Twilio assessments of their postoperative dysuria, urgency and urgency urinary incontinence (as defined above) until it has resolved and remained symptom free x 3 consecutive days. Follow up Twilio assessments at 1month, 3month and 6months will be performed. Patients will concurrently follow up for standard postoperative face-to-face or virtual visit evaluations with their surgical team at 3months.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo HoLEP for bladder outlet obstruction due to the prostate.
* Able to give informed consent.
* Age 18 years or older.

Exclusion Criteria:

* Inability to give informed consent.
* Age less than 18 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patient reported postoperative UUI | 1 month
  Rate of patient reported postoperative UUI

SECONDARY OUTCOMES:
AE reported via Clavien-Dindo classification | 24 hours
  AE reported via Clavien-Dindo classification
Time from HoLEP to postoperative dysuria resolution | 90 days
  Time from HoLEP to postoperative dysuria resolution
Time from HoLEP to postoperative urgency resolution | 90 days
  Time from HoLEP to postoperative urgency resolution
Enucleation/Operative time | 24 hours
  Enucleation/Operative time
Total laser energy used | 24 hours
  Total laser energy used
Perioperative change in hemoglobin | 6 months
  Perioperative change in hemoglobin
Laser repair/maintenance rates | 1 year
  Laser repair/maintenance rates
New postoperative urgency incontinence rates at 1month, 3months and 6months. | 6 months
  New postoperative urgency incontinence rates at 1month, 3months and 6months.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelino Rivera, MD, Principal Investigator — IU Health Physicians
Locations (1):
- IU Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry SJ, Coffey DS, Walsh PC, Ewing LL. The development of human benign prostatic hyperplasia with age. J Urol. 1984 Sep;132(3):474-9. doi: 10.1016/s0022-5347(17)49698-4. PMID 6206240
- [Background] Gilling PJ, Kennett K, Das AK, Thompson D, Fraundorfer MR. Holmium laser enucleation of the prostate (HoLEP) combined with transurethral tissue morcellation: an update on the early clinical experience. J Endourol. 1998 Oct;12(5):457-9. doi: 10.1089/end.1998.12.457. PMID 9847070
- [Background] Tan AH, Gilling PJ, Kennett KM, Frampton C, Westenberg AM, Fraundorfer MR. A randomized trial comparing holmium laser enucleation of the prostate with transurethral resection of the prostate for the treatment of bladder outlet obstruction secondary to benign prostatic hyperplasia in large glands (40 to 200 grams). J Urol. 2003 Oct;170(4 Pt 1):1270-4. doi: 10.1097/01.ju.0000086948.55973.00. PMID 14501739
- [Background] Tan A, Liao C, Mo Z, Cao Y. Meta-analysis of holmium laser enucleation versus transurethral resection of the prostate for symptomatic prostatic obstruction. Br J Surg. 2007 Oct;94(10):1201-8. doi: 10.1002/bjs.5916. PMID 17729384
- [Background] McVary KT, Roehrborn CG, Avins AL, Barry MJ, Bruskewitz RC, Donnell RF, Foster HE Jr, Gonzalez CM, Kaplan SA, Penson DF, Ulchaker JC, Wei JT. Update on AUA guideline on the management of benign prostatic hyperplasia. J Urol. 2011 May;185(5):1793-803. doi: 10.1016/j.juro.2011.01.074. Epub 2011 Mar 21. PMID 21420124
- [Background] Salonia A, Suardi N, Naspro R, Mazzoccoli B, Zanni G, Gallina A, Bua L, Scattoni V, Rigatti P, Montorsi F. Holmium laser enucleation versus open prostatectomy for benign prostatic hyperplasia: an inpatient cost analysis. Urology. 2006 Aug;68(2):302-6. doi: 10.1016/j.urology.2006.02.007. PMID 16904441
- [Background] Elhilali MM, Badaan S, Ibrahim A, Andonian S. Use of the Moses Technology to Improve Holmium Laser Lithotripsy Outcomes: A Preclinical Study. J Endourol. 2017 Jun;31(6):598-604. doi: 10.1089/end.2017.0050. Epub 2017 Apr 25. PMID 28340540
- [Background] Large T, Nottingham C, Stoughton C, Williams J Jr, Krambeck A. Comparative Study of Holmium Laser Enucleation of the Prostate With MOSES Enabled Pulsed Laser Modulation. Urology. 2020 Feb;136:196-201. doi: 10.1016/j.urology.2019.11.029. Epub 2019 Nov 30. PMID 31790785
- [Background] Houssin V, Olivier J, Brenier M, Pierache A, Laniado M, Mouton M, Theveniaud PE, Baumert H, Mallet R, Marquette T, Villers A, Robert G, Rizk J. Predictive factors of urinary incontinence after holmium laser enucleation of the prostate: a multicentric evaluation. World J Urol. 2021 Jan;39(1):143-148. doi: 10.1007/s00345-020-03169-0. Epub 2020 Mar 26. PMID 32219512
- [Background] Kobayashi S, Yano M, Nakayama T, Kitahara S. Predictive risk factors of postoperative urinary incontinence following holmium laser enucleation of the prostate during the initial learning period. Int Braz J Urol. 2016 Jul-Aug;42(4):740-6. doi: 10.1590/S1677-5538.IBJU.2015.0477. PMID 27564285
- [Background] Hur WS, Kim JC, Kim HS, Koh JS, Kim SH, Kim HW, Cho SY, Cho KJ. Predictors of urgency improvement after Holmium laser enucleation of the prostate in men with benign prostatic hyperplasia. Investig Clin Urol. 2016 Nov;57(6):431-436. doi: 10.4111/icu.2016.57.6.431. Epub 2016 Oct 24. PMID 27847917
- [Background] Becker B, Gross AJ, Netsch C. Safety and efficacy using a low-powered holmium laser for enucleation of the prostate (HoLEP): 12-month results from a prospective low-power HoLEP series. World J Urol. 2018 Mar;36(3):441-447. doi: 10.1007/s00345-017-2159-5. Epub 2017 Dec 23. PMID 29275506
- [Background] Elshal AM, El-Nahas AR, Ghazy M, Nabeeh H, Laymon M, Soltan M, Ghobrial FK, El-Kappany HA. Low-Power Vs High-Power Holmium Laser Enucleation of the Prostate: Critical Assessment through Randomized Trial. Urology. 2018 Nov;121:58-65. doi: 10.1016/j.urology.2018.07.010. Epub 2018 Jul 19. PMID 30031005
- [Background] Stern KL, McAdams SB, Cha SS, Abdul-Muhsin HM, Humphreys MR. A New Laser Platform for Holmium Laser Enucleation of the Prostate: Does the Lumenis Pulse 120H Laser Platform Improve Enucleation Efficiency? Urology. 2017 Apr;102:198-201. doi: 10.1016/j.urology.2016.12.022. Epub 2016 Dec 23. PMID 28017884
- [Background] Rivera ME, Lingeman JE, Krambeck AE. Holmium Laser Enucleation of the Prostate. J Endourol. 2018 May;32(S1):S7-S9. doi: 10.1089/end.2017.0710. PMID 29774816